CLINICAL TRIAL: NCT03330002
Title: Post-Market Clinical Registry to Evaluate the Safety and Performance of MANTA Vascular Closure Device (VCD) Under Real World Conditions in the European Union (EU)
Brief Title: MANTA Registry for Vascular Large-bore Closure
Acronym: MARVEL
Status: Completed | Type: Observational
Sponsor: Essential Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PSD-212
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Femoral Arteriotomy Closure
Keywords: Arterial Closure Device; Large Bore Closure Device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- CE-marked MANTA vascular closure devices per IFU: Transcatheter Aortic Valve Replacement (TAVR), Endovascular aneurysm repair (EVAR), TEVAR, etc.
  Interventions: Device: CE-marked MANTA vascular closure device (VCD)

INTERVENTIONS:
Device: CE-marked MANTA vascular closure device (VCD) — Compile real word data on MANTA VCD.

SUMMARY:
The aim of this observational post market study is to compile real world outcome data on the use of the Conformité Européenne (CE) marked MANTA Vascular Closure Device following percutaneous cardiac or peripheral procedures for large bore (10-18F ID) interventional devices.

ELIGIBILITY:
Per MANTA VCD Instructions for Use (IFU)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing percutaneous cardiac or peripheral procedures for large bore (10-18F ID) interventional devices.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Van Mieghem, MD, Principal Investigator — Erasmus Medical Center Rotterdam Netherlands
Locations (9):
- Canada (2):
  - St Paul's Hospital, Vancouver
  - Vancouver General Health, Vancouver
- Aarhus University Hospital, Aarhus, Denmark
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - University of Turku, Turku
- Netherlands (3):
  - OLVG, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Erasmus Medical Center, Rotterdam
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided

REFERENCES:
- [Background] Kadakia MB, Herrmann HC, Desai ND, Fox Z, Ogbara J, Anwaruddin S, Jagasia D, Bavaria JE, Szeto WY, Vallabhajosyula P, Li R, Menon R, Kobrin DM, Giri J. Factors associated with vascular complications in patients undergoing balloon-expandable transfemoral transcatheter aortic valve replacement via open versus percutaneous approaches. Circ Cardiovasc Interv. 2014 Aug;7(4):570-6. doi: 10.1161/CIRCINTERVENTIONS.113.001030. Epub 2014 Jul 15. PMID 25027520
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium (VARC)-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document (VARC-2). Eur J Cardiothorac Surg. 2012 Nov;42(5):S45-60. doi: 10.1093/ejcts/ezs533. Epub 2012 Oct 1. PMID 23026738

RESULTS

PARTICIPANT FLOW:
Groups:
- MANTA Vascular Closure Device (VCD): MANTA VCD following percutaneous cardiac or peripheral procedures (TAVI, MCS, EVAR, TEVAR) for large bore (10-18F ID) interventional devices.
Period: Overall Study
Arm/Group | MANTA Vascular Closure Device (VCD)
Started | 500 (Subjects that received the MANTA VCD)
Completed | 478 (Subjects that received the MANTA VCD and completed 30 day follow-up visit)
Not Completed | 22
Not completed — Lost to Follow-up | 15
Not completed — Death | 7

BASELINE CHARACTERISTICS:
Arm/Group | MANTA Vascular Closure Device (VCD)
Number analyzed (Participants) | 500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 491
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226
  Male | 274
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 71
  Netherlands | 277
  Finland | 96
  Denmark | 29
  Switzerland | 27

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis
Description: The elapsed time between MANTA deployment (withdrawal of sheath from artery) and first observed and confirmed arterial hemostasis (no or minimal subcutaneous oozing and the absence of expanding or developing hematoma).
Time Frame: Immediately after deployment of MANTA VCD
Population: Time to Hemostasis (TTH) was captured in 491/500 subject; 9 subjects did not have TTH recorded.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | MANTA Vascular Closure Device (VCD)
Number analyzed (Participants) | 491
seconds | 50 [20 to 120]

2. Primary Outcome: Number of Participants With One or More Major Access Site Related Complications
Description: Major access site related complications adapted from the VARC-2 definitions
Time Frame: within 30 days of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | MANTA Vascular Closure Device (VCD)
Number analyzed (Participants) | 500
Participants | 20

3. Secondary Outcome: Number of Participants With One or More Minor Access Site Related Complications
Description: Minor access site related complications adapted from the VARC-2 definitions
Time Frame: within 30 days of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | MANTA Vascular Closure Device (VCD)
Number analyzed (Participants) | 500
Participants | 29

ADVERSE EVENTS:
Time Frame: Approximately 30 days after deployment of the MANTA device
Arm/Group | MANTA Vascular Closure Device (VCD)
All-Cause Mortality (participants affected / at risk) | 7/500
Serious Adverse Events (participants affected / at risk) | 110/500
Other Adverse Events (participants affected / at risk) | 98/500
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MANTA Vascular Closure Device (VCD) (N=500)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 2 (2)
Bundle branch block left (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 5 (5)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 4 (4)
Paravalvular aortic regurgitation (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Melaena (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Device embolisation (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vascular access site infection (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 6 (6)
Vascular access site bleeding-oozing (Injury, poisoning and procedural complications) | 17 (17)
Vascular access site occlusion (Injury, poisoning and procedural complications) | 5 (5)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 5 (5)
Haemoglobin decreased (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 15 (15)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 3 (3)
Lead dislodgement (Product Issues) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 36 (36)
Iliac artery perforation (Vascular disorders) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 3 (3)
Peripheral artery stenosis (Vascular disorders) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
Peripheral embolism (Vascular disorders) | 2 (2)
Vessel perforation (Vascular disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MANTA Vascular Closure Device (VCD) (N=500)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 38 (38)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 70 (70)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Institution and Principal Investigator agree that they shall not, without the Sponsor's prior written consent, independently Publish any results of or information about the activities conducted until the multicenter publication is released. If a multi-center manuscript is not submitted for publication within one (1) year after completion of the multi-center Study, Research Institution and Principal Investigator shall have the right to Publish results.

DOCUMENTS (2):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT03330002/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT03330002/SAP_001.pdf